CLINICAL TRIAL: NCT01975415
Title: Digital Medicine in Meditation
Acronym: DigMed2
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: The Chopra Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13 - 6251
Record Dates: First submitted 2013-10-17; First posted 2013-11-04 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Biometric Changes During Meditation
Keywords: Meditation; Sensors; Digital medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experienced Meditators: Self-identified participants who confirm to having a regular meditation practice for at least 3 months and practiced at least 70 minutes per week.
- Novice meditators: Self-identified participant who confirm to either having never seriously tried meditation, or who have not meditated more than once a week for at least 3 months

SUMMARY:
This study will investigate the acute response to meditation during a week-long meditation retreat at the Chopra Center as measured by the continuous, simultaneous monitoring of numerous biometric parameters in selected cohorts of experienced and novice meditators during periods of meditation and specific breathing techniques. Comparisons between cohorts as well as over time will allow for the identification of meditation and/or breathing-related changes.

DETAILED DESCRIPTION:
The biometric responses to meditation and breathing techniques will be compared between novice and experienced meditators, as well as initial versus final biometric responses in all participants stratified by cohort. Investigators hypothesize that novice meditators will experience a measurable change in response to mediation over the week-long retreat, whereas experienced meditators will demonstrate a more robust response than novice meditators on the first day of the retreat with less change over the retreat.

ELIGIBILITY:
Inclusion Criteria:

* Adult over age 18 who are already registered to participate in the week-long "Seduction of the Soul" retreat.
* Capable of providing informed consent

Exclusion Criteria:

* Chronic requirement for daily use of chronotropically active medications including beta-blockers, non-dihydropyridine calcium channel blockers, clonidine or beta-agonist inhalers.
* Implantable pacemaker or cardioverter-defibrillator.
* Known allergy to adhesives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be a subset of 40 individuals from a total of ~200 who self-selected to participate in a week-long "Seduction of Spirit" retreat at The Chopra Center in the La Costa Resort in Carlsbad, CA. The 40 anticipated participants will be made up of 2 cohorts: experienced meditators and novice meditators.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Participants will be measured at Day 1 and Day 5 of retreat
  Non-invasive blood pressure
ECG | Participants will be measured at Day 1 and Day 5 of retreat
  5-lead electrocardiogram
Respiration rate | Participants will be measured at Day 1 and Day 5 of retreat
  Respiration rate
Heart Rate | Participants will be measured at Day 1 and Day 5 of retreat
  Heart rate
Oxygen saturation (SpO2) | Participants will be measured at Day 1 and Day 5 of retreat
  Oxygen saturation
Skin temperature | Participants will be measured at Day 1 and Day 5 of retreat
  Skin temperature
Heart rate variability | Participants will be measured at Day 1 and Day 5 of retreat
  Variability in heart rate across a period of time.
EEG | Participants will be measured at Day 1 and Day 5 of retreat
  14-lead Electroencephalogram
Stress level | Participants will be measured at Day 1 and Day 5 of retreat
  Stress level calculated from heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- The Chopra Center, Carlsbad, California, United States